CLINICAL TRIAL: NCT02369016
Title: A Randomized, Double-blind Phase III Study of Copanlisib Versus Placebo in Patients With Rituximab-refractory Indolent Non-Hodgkin's Lymphoma (iNHL) - CHRONOS-2
Brief Title: Phase III Copanlisib in Rituximab-refractory iNHL
Acronym: CHRONOS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17322; 2014-000925-19 (EudraCT Number)
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: indolent Non-Hodgkin lymphoma; rituximab-refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib (BAY 80-6946) (Experimental): patients with rituximab-refractory iNHL
  Interventions: Drug: Copanlisib (BAY 80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY 80-6946) — 60 mg of experimental drug in solution administered intravenously on Days 1, 8 and 15 of each 28-day treatment cycle

SUMMARY:
To assess the safety of copanlisib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of indolent B-cell NHL, with histological subtype limited to the following:

  * Follicular lymphoma (FL) grade 1-2-3a.
  * Small lymphocytic lymphoma (SLL) with absolute lymphocyte count < 5 x 10*9/L at the time of diagnosis and at study entry.
  * Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM).
  * Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal).
* Patients must have received two or more prior lines of treatment. A previous regimen is defined as one of the following: at least two months of single-agent therapy, at least two consecutive cycles of polychemotherapy, autologous transplant, radioimmunotherapy.
* Prior therapy must include rituximab and alkylating agents.Prior exposure to idelalisib or other PI3K inhibitors is acceptable (except to copanlisib) provided that there is no resistance.
* Patients must be refractory to the last rituximab-based treatment, defined as no response or response lasting < 6 months after completion of treatment. Time interval to assess refractoriness will be calculated between the end date (last day) of the last rituximab-containing regimen and the day of diagnosis confirmation of the subsequent relapse.
* Patients must have at least one bi-dimensionally measurable lesion (which has not been previously irradiated) according to the Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.
* Patients affected by WM, who do not have at least one bi-dimensionally measurable lesion in the baseline radiologic assessment, must have measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level ≥ 2 x upper limit of normal (ULN)and positive immunofixation test.
* ECOG performance status ≤ 1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Histologically confirmed diagnosis of FL grade 3b.
* Chronic lymphocytic leukemia (CLL).
* Transformed disease (assessed by investigator):

  * histological confirmation of transformation, or
  * clinical and laboratory signs: rapid disease progression, high standardized uptake value (SUV) (> 12) by positron emission tomography (PET) at baseline if PET scans are performed (optional).
* Bulky disease - Lymph nodes or tumor mass (except spleen) >= 7cm LD (longest diameter)
* Known lymphomatous involvement of the central nervous system.
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's assessment).
* Type I or II diabetes mellitus with HbA1c > 8.5% at Screening.
* Known history of human immunodeficiency virus (HIV) infection.
* Active clinically serious infections > CTCAE Grade 2
* Active Hepatitis B or hepatitis C
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* History of having received an allogeneic bone marrow or organ transplant
* Positive cytomegalovirus (CMV) PCR test at baseline
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Brazil (3):
  - Jaú, São Paulo
  - São Paulo, São Paulo
  - São Paulo
- Plovdiv, Bulgaria
- Athens, Greece
- Italy (2):
  - Bologna, Emilia-Romagna
  - Genoa, Liguria
- Gdynia, Poland
- Russia (5):
  - Kazan'
  - Kemerovo
  - Moscow
  - Omsk
  - Penza
- Johannesburg, Gauteng, South Africa
- South Korea (4):
  - Seoul, Seoul Teugbyeolsi
  - Jeollabuk-do
  - Jeollanam-do
  - Seoul
- Taipei, Taiwan
- Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 study centers in 10 countries/regions: Brazil (2), Bulgaria (1), Greece (1), Italy (2), Poland (1), Russian Federation (5), South Africa (1), South Korea (5), Taiwan (1) and Turkey (1) between 22 September 2015 (first patient first visit) and 26 October 2022 (last patient last visit).
Pre-assignment Details: 34 participants were screened. 9 participants were screening failures and 25 participants were randomized to study treatment: 17 to copanlisib and 8 to placebo. All randomized participants also received at least one dose of study treatment and were valid for safety analyses. After study unblinding 7 placebo participants switched to copanlisib.
Groups:
- Copanlisib (BAY80-6946, Aliqopa): Participants who were randomized to copanlisib until end of the study
- Placebo: Participants who were randomized to placebo until switching from placebo to copanlsib after disease progression or after study unblinding
Period: Overall Study
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo
Started | 17 | 8
Switched to Copanlisib After Study Unblinding | 0 | 7
Completed | 0 | 0
Not Completed | 17 | 8
Not completed — AE associated with clinical disease progression | 2 | 1
Not completed — AE not associated with clinical diseaseprogression | 4 | 1
Not completed — Progressive disease - clinical progression | 1 | 4
Not completed — withdrawal by patient | 4 | 0
Not completed — Progressive disease - radiological progression | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants who were randomized to placebo until switching from placebo to copanlisib after disease progression or after study unblinding
- Total: Total of all reporting groups
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 12 | 5 | 17
  From 65-84 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)s
Description: Adverse event data were collected after signing the informed consent until 30 days after the last study drug administration (end of safety follow-up)
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Groups:
- Switched to Copanlisib: Participants who switched from placebo to copanlisib
- Treated With Copanlisib: Participants who were treated with copanlisib (randomized to copanlisib + switched from placebo to copanlisib)
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo | Switched to Copanlisib | Treated With Copanlisib
Number analyzed (Participants) | 17 | 8 | 7 | 24
Participants | 17 | 7 | 7 | 24

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAE)s
Description: Serious adverse event data were collected after signing the informed consent until 30 days after the last study drug administration (end of safety follow-up)
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Patients who were randomized to placebo until switching from placebo to copanlsib after disease progression or after study unblinding
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo | Switched to Copanlisib | Treated With Copanlisib
Number analyzed (Participants) | 17 | 8 | 7 | 24
Participants | 6 | 1 | 5 | 11

3. Primary Outcome: Number of Participants With Abnormal Laboratory Parameters
Description: - Above threshold of 10% and reported as TEAEs - any event (Grade 1-4)
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo | Switched to Copanlisib | Treated With Copanlisib
Number analyzed (Participants) | 17 | 8 | 7 | 24
Participants
  ANY | 9 | 1 | 3 | 12
  Hyperglycaemia | 6 | 0 | 4 | 10
  Neutropenia | 6 | 0 | 1 | 7
  Neutrophil count decreased | 4 | 0 | 2 | 6
  Anaemia | 2 | 2 | 4 | 6
  Platelet count decreased | 3 | 0 | 2 | 5

4. Primary Outcome: Number of Participants With Abnormal Vital Signs
Description: - Reported as TEAEs - worst CTCAE grade total -
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib (BAY80-6946, Aliqopa) | Placebo | Switched to Copanlisib | Treated With Copanlisib
Number analyzed (Participants) | 17 | 8 | 7 | 24
Participants
  Blood pressure increased | 2 | 0 | 1 | 3
  Electrocardiogram QT prolonged | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: from the start of study drug administration until 30 days after the last study drug administraion, up to end of safety follow-up, approximately 7 years
Groups:
- Randomized to Copanlisib: Participants who were randomized to copanlisib until end of the study
- Randomized to Placebo: Participants who were randomized to placebo until switching from placebo to copanlsib after disease progression or after study unblinding
Arm/Group | Randomized to Copanlisib | Randomized to Placebo | Switched to Copanlisib | Treated With Copanlisib
All-Cause Mortality (participants affected / at risk) | 2/17 | 1/8 | 2/7 | 4/24
Serious Adverse Events (participants affected / at risk) | 6/17 | 1/8 | 5/7 | 11/24
Other Adverse Events (participants affected / at risk) | 17/17 | 7/8 | 7/7 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Copanlisib (N=17) | Randomized to Placebo (N=8) | Switched to Copanlisib (N=7) | Treated With Copanlisib (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Copanlisib (N=17) | Randomized to Placebo (N=8) | Switched to Copanlisib (N=7) | Treated With Copanlisib (N=24)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (11) | 6 (13)
Lymphopenia (Blood and lymphatic system disorders) | 1 (11) | 0 (0) | 0 (0) | 1 (11)
Neutropenia (Blood and lymphatic system disorders) | 6 (14) | 0 (0) | 1 (4) | 7 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (6) | 1 (3) | 1 (3)
Conjunctivitis allergic (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (12) | 0 (0) | 1 (6) | 4 (18)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 3 (5) | 0 (0) | 2 (2) | 5 (7)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6) | 1 (1) | 0 (0) | 2 (6)
Fatigue (General disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (4)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (6) | 0 (0) | 3 (4) | 5 (10)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immunodeficiency common variable (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (2) | 2 (5)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 4 (5)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (12) | 0 (0) | 1 (7) | 3 (19)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (9) | 0 (0) | 2 (4) | 6 (13)
Platelet count decreased (Investigations) | 3 (5) | 0 (0) | 2 (4) | 5 (9)
Weight decreased (Investigations) | 2 (4) | 1 (1) | 1 (1) | 3 (5)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (107) | 0 (0) | 4 (59) | 10 (166)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 4 (6)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (8) | 1 (1) | 0 (0) | 3 (8)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (4) | 5 (7)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 2 (3) | 1 (1) | 2 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (32) | 1 (1) | 2 (19) | 5 (51)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02369016/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02369016/SAP_001.pdf